CLINICAL TRIAL: NCT07307911
Title: Neuroprotective Effects of Coenzyme Q10 in Paclitaxel-Induced Peripheral Neuropathy
Brief Title: Coenzyme Q10 for Neuroprotection in Paclitaxel-Induced Neuropathy
Acronym: Co-Pa-N
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CoQ10-PN-2025-01
Record Dates: First submitted 2025-12-04; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — coenzyme Q10; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoQ10 group (Experimental): Participants in this arm will receive standard weekly paclitaxel chemotherapy (80 mg/m²) for twelve weeks in combination with Coenzyme Q10 supplementation at 200 mg twice daily. The purpose of this arm is to evaluate the effect of Coenzyme Q10 on chemotherapy-induced peripheral neuropathy, fatigue, pain, and related serum biomarkers.
  Interventions: Dietary Supplement: Coenzyme Q 10; Drug: Paclitaxel
- Control group (Placebo Comparator): Participants in this arm will receive standard weekly paclitaxel chemotherapy (80 mg/m²) for twelve weeks without Coenzyme Q10 supplementation. This arm serves as a comparator to evaluate the effects of Coenzyme Q10 on chemotherapy-induced peripheral neuropathy, fatigue, pain, and related serum biomarkers.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Dietary Supplement: Coenzyme Q 10 — Coenzyme Q10 200 mg orally twice daily for twelve weeks, for CoQ 10 grpup only
  Arms: CoQ10 group
Drug: Paclitaxel — : Paclitaxel 80 mg/m² administered weekly for twelve weeks to Control and CoQ groups

SUMMARY:
* This study aims to investigate whether Coenzyme Q10 supplementation can reduce chemotherapy-induced peripheral neuropathy, fatigue, and pain in women with newly diagnosed breast cancer receiving paclitaxel treatment. The study will also examine the effects of Coenzyme Q10 on biomarkers associated with nerve damage. The main questions it seeks to answer are:
* Does Coenzyme Q10 improve patients' quality of life by reducing neuropathy, fatigue, and pain during chemotherapy?
* How does Coenzyme Q10 affect serum levels of nerve growth factor, neurofilament light chain, malondialdehyde, and osteopontin during treatment?
* Participants will: Receive either Coenzyme Q10 along with standard weekly paclitaxel chemotherapy or paclitaxel alone for twelve weeks.
* Complete questionnaires on neuropathy, fatigue, and pain at the end of each chemotherapy cycle.
* Provide blood samples at the beginning and end of the study to measure biomarkers of nerve injury.

DETAILED DESCRIPTION:
Fifty female patients with newly diagnosed breast cancer scheduled for weekly paclitaxel chemotherapy (80 mg/m2) will be randomized in a 1:1 ratio into two study arms. The CoQ10 Group will receive Coenzyme Q10 supplementation (200 mg twice daily) for twelve weeks in addition to the standard chemotherapy protocol, while the Control Group will receive the standard chemotherapy protocol alone.

Clinical assessments for peripheral neuropathy, including grading via NCI-CTCAE v5.0, will be conducted prior to the initiation of each weekly paclitaxel session to monitor for symptom onset and severity. Patient-reported outcome measures for neuropathy-specific quality of life (FACT/GOG-Ntx12), fatigue (FACIT-F), and pain intensity (VAS) will be administered at baseline and at the end of weeks 3, 6, 9, and 12. To specifically assess pain interference and severity over time, the Brief Pain Inventory (BPI) will be administered at week 6 and week 12.

For the exploratory biomarker analysis, 5 mL of venous blood will be collected via antecubital venipuncture at baseline (one hour before the first cycle) and one hour after the final paclitaxel dose. Samples will be allowed to clot at room temperature for 30 minutes, then centrifuged at 3,000 rpm for 15 minutes. The resulting serum will be aliquoted and stored at -80 degrees Celsius. Biochemical quantification of NGF, NfL, and OPN will be performed using double-antibody sandwich ELISA, and MDA levels will be determined via colorimetric assay to evaluate oxidative stress and axonal integrity. All participants will be followed for a total of 90 days from the start of treatment to evaluate the time to development of Grade 2 or 3 neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older with newly diagnosed breast cancer.
* Chemotherapy-naïve (have not received prior chemotherapy).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Severe cardiovascular disease (left ventricular ejection fraction <55%).
* Hereditary muscle disorders.
* Diabetes mellitus or history of alcoholism.
* Thyroid dysfunction.
* History of allergy to Coenzyme Q10 or related compounds.
* Advanced liver disease (liver enzyme elevation >3× upper limit of normal or cirrhosis).
* Chronic kidney disease (CKD), defined as estimated glomerular filtration rate <60 mL/min/m².

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Paclitaxel-Induced Peripheral Neuropathy | From baseline to the end of four chemotherapy cycles (approximately 12 weeks)
  The occurrence of peripheral neuropathy in patients receiving paclitaxel chemotherapy will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4. This will evaluate the onset and severity of neuropathy symptoms, including numbness, tingling, and pain in hands and feet.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity 12-item questionnaire (FACT/GOG-Ntx12) | Baseline, week 3, week 6, week 9, and week 12.
  A 12-item questionnaire used to assess the impact of peripheral neuropathy on daily functioning. Each item is scored from 0 ("not at all") to 4 ("very much"). The total score is calculated by multiplying the sum of individual item scores by 12 and dividing by the number of items completed. Scores range from 0 to 48. Higher scores indicate better neuropathy-related quality of life.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Baseline, week 3, week 6, week 9, and week 12.
  A 13-item scale evaluating fatigue severity. Each item is scored on a 0-4 Likert scale. Total scores are calculated by summing individual item scores, multiplying by 13, and dividing by the number of items completed. Scores range from 0 to 52. Higher FACIT-F scores indicate less fatigue and better quality of life.
Visual Analog Scale (VAS) for Pain | Baseline, week 3, week 6, week 9, and week 12.
  A 100-mm horizontal line used to assess neuropathic pain at rest. The measurement is converted to a 0-10 numeric score, where 0 = "no pain" and 10 = "pain as bad as you can imagine." Higher scores indicate greater pain severity.
Brief Pain Inventory (BPI)-Short Form | Week 6 and week 12.
  The BPI assesses pain severity (4 items) and interference with daily activities (7 items). Each item is rated on a 0-10 scale. A total pain severity score is calculated by averaging the severity items, and an interference score is calculated by averaging the interference items. Scores range from 0 to 10. Higher scores indicate greater pain intensity and interference with daily life.

OTHER OUTCOMES:
Change from Baseline in Serum Nerve Growth Factor (NGF) Levels | Baseline (1 hour before first cycle) and End of Treatment (1 hour after final cycle, approximately Week 12).
  Serum NGF levels will be quantified using a double-antibody sandwich ELISA kit to assess neurotrophic status.Unit of Measure: picograms per milliliter (pg/mL).Higher levels are generally associated with nerve repair/regeneration
Change from Baseline in Serum Neurofilament Light Chain (NfL) Levels | Baseline (1 hour before first cycle) and End of Treatment (1 hour after final cycle, approximately Week 12).
  Serum NfL levels will be measured via ELISA as a biomarker of axonal injury and neurodegeneration.Unit of Measure: picograms per milliliter (pg/mL).Higher levels indicate greater degrees of neuronal damage."
Change from Baseline in Serum Osteopontin (OPN) Levels | Baseline (1 hour before first cycle) and End of Treatment (1 hour after final cycle, approximately Week 12).
  Serum OPN levels will be quantified using a double-antibody sandwich ELISA kit.Unit of Measure: nanograms per milliliter (ng/mL).low OPN is linked to worse neuropathy.
Change from Baseline in Serum Malondialdehyde (MDA) Levels | Baseline (1 hour before first cycle) and End of Treatment (1 hour after final cycle, approximately Week 12).
  MDA will be measured as a marker of lipid peroxidation and oxidative stress using a colorimetric assay kit.Unit of Measure: nanomoles per milliliter (nmol/mL).Higher levels indicate increased oxidative stress."

CONTACTS AND LOCATIONS:
Locations (1):
- Damanhur Oncology Center, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: No